CLINICAL TRIAL: NCT04486651
Title: A Randomized, Double-blinded, Multicenter, Phase III Clinical Study of HX008 (Recombinant Humanized Anti-PD-1 Monoclonal Antibody Injection) Plus Irinotecan Versus Placebo Plus Irinotecan as Second-line Treatment in Advanced Gastric Cancer
Brief Title: HX008 Plus Irinotecan Versus Placebo Plus Irinotecan as Second-line Treatment in Advanced Gastric Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taizhou Hanzhong biomedical co. LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HX008-III-GC-01
Record Dates: First submitted 2020-07-22; First posted 2020-07-24 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Stomach Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Irinotecan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HX008 plus Irinotecan (Experimental): Participants recieve HX008 200 mg intravenous (IV) every 3 weeks (Q3W) plus irinotecan 160 mg/m², IV, Q2W.
  Interventions: Drug: Irinotecan Hydrochloride Injection; Drug: HX008
- Placebo plus Irinotecan (Placebo Comparator): Participants recieve placebo intravenous (IV) every 3 weeks (Q3W) plus irinotecan 160 mg/m², IV, Q2W.
  Interventions: Drug: Irinotecan Hydrochloride Injection; Drug: Placebo

INTERVENTIONS:
Drug: Irinotecan Hydrochloride Injection — 160 mg/m² administered as IV infusion on Day 1 of each 14-day cycle.
Drug: HX008 — 200 mg administered as IV infusion on Day 1 of each 21-day cycle.
  Arms: HX008 plus Irinotecan
Drug: Placebo — Administered as IV infusion on Day 1 of each 21-day cycle.
  Arms: Placebo plus Irinotecan

SUMMARY:
This is a randomized, double-blinded, multicenter study to evaluate the efficacy and safety of HX008 injection combined with irinotecan versus placebo combined with irinotecan as second-line therapy in patients with adcanced gastric or gastroesophageal junction (GEJ) adenocarcinoma who have had tumor progression after first-line treatment with platinum and/or fluropyrimidine therapy.

ELIGIBILITY:
Inclusion Criteria:

* Understood and signed an informed consent form.
* Age ≥ 18 and ≤ 75 years old, male or female.
* Has histologically- or cytologically-confirmed diagnosis of locally advanced unresectable or metastatic adenocarcinoma of stomach or the esophagogastric junction (GEJ).
* Has experienced documented objective radiographic or clinical disease progression during or after first-line therapy containing platinum and/or fluoropyrimidine therapy.
* Willing to provide tissue for PD-L1 biomarker analysis.
* Has a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Score.
* Life expectancy ≥ 3 months.
* Has adequate organ function.
* Female participants of childbearing potential should have a negative pregnancy within 72 hours before the randomization. Male and female participants should agree to use an adequate method of contraception during the experiment and 1 year after the last administration of the test drugs.

Exclusion Criteria:

* Has squamous cell or undifferentiated gastric cancer.
* Diagnosed additional maliganancy within 3 years prior to randomization with the expection of curatively treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin,curatively resected in situ cervival or non-muscle invasive bladder cancers.
* Has had a prior anti-cancer monoclonal antibody within 4 weeks prior to the first dose of trial treatment or who has not recovered (≤ Grade 1 or at Baseline) from AEs due to agents administered more than 4 weeks earlier.
* Has had prior chemotherapy,radiation therapy or targeted small molecular therapy within 2 weeks prior to the first dose of trial treatment or who has not recovered (≤ Grade 1 or at Baseline) from AEs due to a previously administrated agent.
* Has received prior therapy with an anti-PD-1, or anti-PD-L1, or anti-CTLA-4 agents.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Has uncontrolled ascites, pleural effusion, or pericardial effusion.
* Has active autoimmune disease that has required systemic treatment in past 2 years.
* Has received a major surgery within 4 weeks prior to randomization.
* Has received system treatment with corticosteroids (dose >10mg/day prednison or other therapeutic hormones) within 2 weeks prior to the first dose of trial treatment.
* Has incomplete intestinal obstruction, active gastrointestinal hemorrhage and perforation.
* Has a history of non-infectious pneumonitis that required steriods or has current pneumonitis.
* Has any serious and/or uncontrolled disease.
* Has active viral infection.
* Has received a live vaccine within 30 days prior to the first dose of trial treatment.
* Has participated in other anticancer drug clinical trials within 4 weeks.
* According to the judgement of the investigators, there are other factors that may lead to the termination of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560 (Estimated)
Dates: Start 2020-09-16 (Actual); Primary Completion 2023-08-10 (Estimated); Study Completion 2023-08-10 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) in All Participants | Up to approximately 36 months
  OS was defined as the time from randomization to death due to any cause. Participants without documented death at the time of the final analysis were censored at the date of the last follow-up. OS is reported here for all participants in the experimental arm and placebo comparator arm.
Overall Survival (OS) in Participants With PD-L1 CPS≥1 | Up to approximately 36 months
  OS was defined as the time from randomization to death due to any cause. Participants without documented death at the time of the final analysis were censored at the date of the last follow-up. OS is reported here for all participants in the experimental arm and placebo comparator arm with PD-L1 CPS≥1.

SECONDARY OUTCOMES:
Progression-free Survival (PFS) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) | Up to approximately 36 months
  PFS was defined as the time from randomization to the first documented disease progression per RECIST 1.1 assessed by investigators or death due to any cause, whichever occurs first.
Objective Response Rate (ORR) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) | Up to approximately 36 months
  ORR was defined as the percentage of participants who have a complete response (CR) or a partial response (PR), per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as assessed by investigators.
Disease Control Rate (DCR) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) | Up to approximately 36 months
  DCR was defined as the percentage of participants who have a CR or a PR or a stable disease (SD), per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as assessed by investigators.
Duration of Response (DOR) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) | Up to approximately 36 months
  DOR was defined as the time from the first documented evidence of a response of CR or PR, per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as assessed by investigators.

CONTACTS AND LOCATIONS:
Locations (64):
- China (64):
  - Anhui Provincial Cancer Hospital, Hefei, Anhui
  - Anhui Provincial Hospital, Hefei, Anhui
  - The Second Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing ChaoYang Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Peking University Internationale Hospital, Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Xiamen, Fujian
  - Gansu Wuwei Tumor Hospital, Wuwei, Gansu
  - Affiliated Cancer Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Zhongshan People's Hospital, Guangzhou, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - Cancer Hospital Chinese Academy of Medical Sciences, Shenzhen Center, Shenzhen, Guangdong
  - Guangxi Medical University Cancer Hospital, Naning, Guangxi
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangzhou
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Affiliated Hospital of Hebei University, Shijiazhuang, Hebei
  - The affiliated Cancer Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The First Affiliated Hospital of Henan Science&Technology University, Zhengzhou, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - The Second Xiangya Hospital of Cancer South University, Changsha, Hunan
  - Xiangya Hospital, Central South University, Changsha, Hunan
  - Hunan Cancer Hospital, Changsha, Hunan
  - The Affiliated People's Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - Changzhou Cancer Hospital, Changzhou, Jiangsu
  - Jiangsu Provincial Hospital, Nanjing, Jiangsu
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Zhongda Hospital Southeast Universtiy, Nanjing, Jiangsu
  - Nantong Tumor Hospital, Nantong, Jiangsu
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - Yangzhou FIrst People's Hospital, Yangzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Jiangxi Cancer Hospital, Nanchang, Jiangxi
  - Jilin Cancer Hospital, Changchun, Jilin
  - The First Hospital of Jilin University, Changchun, Jilin
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Liaoning Cancer Hospital, Shenyang, Liaoning
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Shandong Provincial Hospital, Jinan, Shandong
  - Shandong Cancer Hospital, Jinan, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality
  - Shanxi Cancer Hospital, Taiyuan, Shanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - Sichuan Cancer Hospital, Chengdu, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Hubei Cancer Hospital, Hubei, Wuhan
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Xinjiang Medical University Cancer Hospital, Ürümqi, Xinjiang
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital, Medical School of Zhejiang University, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No